CLINICAL TRIAL: NCT02257255
Title: Classic Cesarean Section Versus Minimally Invasive Cesarean Section: Pain Assessment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Vale do Sapucai (Other)
Responsible Party: Principal Investigator, Ivanildo Archangelo Junior, MD, Universidade do Vale do Sapucai
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: cesarean
Record Dates: First submitted 2014-08-18; First posted 2014-10-06 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Pregnancy
Keywords: cesarean section; pain, postoperative/diagnosis; pain measurement/methods
MeSH Terms: conditions — Pain; Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pfannenstiel cesarean section (Active Comparator): Women in 36 to 40 weeks of pregnancy undergoing first cesarean section by Pfannenstiel technique. Pain assessment on postoperative hours 6, 12 and 24.
  Interventions: Procedure: Pfannenstiel cesarean section
- Misgav-Ladach cesarean section (Experimental): Women in 36 to 40 weeks of pregnancy undergoing first cesarean section by minimally invasive technique. Pain assessment on postoperative hours 6, 12 and 24.
  Interventions: Procedure: Misgav-Ladach cesarean section

INTERVENTIONS:
Procedure: Pfannenstiel cesarean section — Pain scales ( VAS and McGill ) 6, 12 and 24 hours after cesarean to pain assessment
  Arms: Pfannenstiel cesarean section
Procedure: Misgav-Ladach cesarean section — Pain scales (VAS and McGill) 6, 12 and 24 hours ater cesarean to pain assessment
  Arms: Misgav-Ladach cesarean section

SUMMARY:
Cesarean section is the most performed abdominal surgery in women, worldwide. The World Health Organization (WHO) considers 15% of deliveries the ideal rate of this surgery. However, Brazil presents the highest rates of cesarian section in the world, reaching 85% in hospitals and private clinics.

The most used technique of cesarean section is the known as Pfannenstiel or Classical technique. In 1996, a new technique was described, called Misgav Ladach or minimally invasive technique.

Several studies have show that the minimally invasive technique is faster and promotes lower costs and less intraoperative bleeding. There is no current evidence that this technique is less painful.

This study aims to compare the postoperative pain in both techniques,by means of two pain scales: a one-dimensional scale, the Visual Analogue Scale, and a multidimensional scale, the McGill Scale.

DETAILED DESCRIPTION:
1. STUDY

   Primary, clinical, prospective, randomized, double blind with, controlled, two parallel groups interventional and analytical.
2. MATERIAL

A-CALCULATION OF SAMPLE SIZE

Were used to calculate the size of the sample study data Antalon et al. (2001), who also compared the two techniques of caesarean section, and the Student's t-test was used bi flow. Considering a standard deviation of 1.5 points in the Visual Analog Pain Scale, and significant a difference of two points, the calculated number of patients per group was 15, with a significance level of 5% and power of 95 test %.

C RANDOMIZATION AND CONFIDENTIALITY OF ALLOCATION

The allocation will be determined by random sequence generated by computer (BioStat 5.0 software, Mamiraua Institute, Brazil). The sequence had been held by the researcher who will make allocation of patients to groups in caesarean Pfannenstiel or Misgav-Ladach, 15 in each group.

D-PROCEDURES

ANESTHESIA:

In both groups will be performed spinal anesthesia at L2-L4 with heavy bupivacaine 13 mg and morphine 0.1 mg% standardized by the Anesthesiology Service of HCSL.

SURGICAL PROCEDURE:

Surgical procedure (classical technique)

Once displayed, according to the behavior of the service, this will be performed according to the following surgical technique:

* Traditional Preparation: pubic shaving, prior bladder emptying.
* Asepsis with degerminate clorhexidine and alcoholic
* The transverse abdominal incision approximately 10 cm, 3-4 cm above the pubic symphysis.
* Cross Opening subcutaneous tissue.
* Opening Aponeurosis transversely, hemostasis of bleeding vessels.
* Separation by dissection of the anterior rectus sheath muscles of the abdomen to the umbilicus.
* Separation of the muscles of the median raphe manually, exposure, clamping and opening the parietal peritoneum with scissors longitudinally.
* Opening of the visceral peritoneum transversely with scissors, taking off the bladder from the uterus.
* Hysterotomy segment transverse, arcuate, superior concavity, made a small incision with a scalpel and that is complete with Kelly forceps to reach the uterine cavity and then enlarging it with fingers without taking off the bladder from the uterus.
* Disposal of amniotic fluid. fetal extraction, using the leverage if necessary.
* Clamping of the umbilical cord and immediate care to the newborn.
* Administration of cefazolin 2g IV and 10 IU oxytocin.
* Afterbirth and revision of the uterine cavity.
* Hysterorrhaphy with Catgut chrome one in a continuous suture not anchored.
* Visceral peritonization simple catgut and 2-0 suture in simple running suture.
* Revision of the abdominal cavity.
* Closure of the parietal peritoneum and with simple catgut 2-0 suture in simple running suture.
* Closing the muscular plane is separated into "U", with simple catgut fioa 2-0 points.
* Closing the aponeurosis chrome catgut sutures in one not anchored.
* Approximation of the subcutaneous tissue with 2-0 catgut simple in separate points.
* Skin closure is made with nylon suture with 4-0 points Donati modified.
* Dressing kept simple in the early hours.

Surgery (minimally invasive technique)

Once displayed, according to the behavior of the service, this will be performed according to the following surgical technique:

* Traditional Preparation: pubic shaving, prior bladder emptying.
* Asepsis and degermante with alcoholic chlorhexidine.
* The transverse abdominal incision approximately 10 cm, 3-4 cm above the pubic symphysis.
* Cross Opening subcutaneous tissue with electrocautery used in clotting.
* Opening Aponeurosis transversely, hemostasis of bleeding vessels.
* Separation of the Muscles of the median raphe manually, exposure, clamping the parietal peritoneum, small opening with scissors. Through digital dilatation peritoneum is opened across the entire length of the incision.
* Hysterotomies Segment transverse, arcuate, superior concavity, made a small incision with a scalpel and that is complete with Kelly forceps to reach the uterine cavity and then enlarging it with fingers without taking off the bladder from the uterus.
* Disposal of amniotic fluid. Fetal extraction, using the leverage if necessary.
* Clamping of the umbilical cord and immediate care to the newborn.
* Administration of cefazolin 1 g IV and 10 IU oxytocin.
* And revision of the uterine cavity.
* Hysterorrhaphy with Catgut chrome one in a continuous suture not anchored.
* Revision of the abdominal cavity.
* Closing the aponeurosis chrome catgut sutures in one not anchored.
* Approximation of the subcutaneous tissue with 2-0 catgut simple in separate points.
* Skin closure is made with nylon suture with 4-0 points Donati modified.
* Dressing kept simple in the early hours]. Postoperative medication
* Intravenous hydration with 1000 ml of glucose 5% and 500 ml of 0.9% saline solution in drip 60 drops / minute.
* Use (dimethicone) every 8 hours the first dose at 12 hours postoperatively.
* Use of analgesic and anti-spasmodic every 6 hours if needed (Buscopan composts® (scopolamine butylbromide 20mg and dipyrone 2.5 mg).

F-STATISTICAL METHOD The data will be tabulated and subjected to statistical analysis. The level of rejection of the null hypothesis will be set at 5% (α <0.05).

For numeric variables will be used descriptive statistics, with calculations of median, mean and deviation padrão.O Mann-Whitney test is used to compare two independent groups with nonparametric behavior and the chi-square test for categorical variables.

ELIGIBILITY:
INCLUSION CRITERIA:

* Primiparous patients who are undergoing cesarean section

EXCLUSION CRITERIA:

* Previous pelvic and/or abdominal surgery ;
* Emergency cesarean section, due to placenta previa, fetal distress, cord prolapse or other obstetric emergencies;
* Pregnancies below 36 weeks.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-05; Primary Completion 2015-02 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Pain | Postoperative 24 hours
  pain assessment using two kinds of pain scales VAS and McGILL scale at 6, 12 and 24 hours of postoperative

SECONDARY OUTCOMES:
time spent in two different techniques for cesarean | 1 hour
  compare time spent in each technique, considering only cesarean that spent less than 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: IVANILDO ARCHANGELO, Principal Investigator — UNIVERSIDADE DO VALE DO SAPUCAÍ; Daniela F Veiga, MD, PhD, Study Chair — Universidade do Vale do Sapucaí
Locations (1):
- Ivanildo Archangelo Jr, Pouso Alegre, Minas Gerais, Brazil